CLINICAL TRIAL: NCT00949923
Title: Green Tea Supplement in Women With Incident Breast Cancer
Brief Title: Green Tea in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1B-08-1; HS-07-00731
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Incident Breast Cancer
Keywords: Postmenopausal women; Suspicious for breast ca
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tea capsules (Active Comparator): 3 tea capsules daily for 3 weeks
  Interventions: Dietary Supplement: tea capsule
- Control (No Intervention): No tea capsules

INTERVENTIONS:
Dietary Supplement: tea capsule — 3 tea capsules daily for 3 weeks
  Other Names: Green Tea Mega EGCG, ProHealth, Inc
  Arms: tea capsules

SUMMARY:
Prognostic factors for breast cancer beyond stage at diagnosis and tumor characteristics have not been well studied. Of special interest are lifestyle factors that can be modified by women after diagnosis to increase disease-free survival. Green tea is rich in polyphenols consisting primarily of epicatechins, epigallocatechin, epicatechin gallate, and epigallocatechin gallate (EGCG). The investigators hypothesize that there will be a reduction in proliferation and/or an increase in apoptosis in association with short-term EGCG treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (at least 2 years since last menstrual period) or age 55 or older if prior hysterectomy
* Non-current (not with past 6 months) user of menopausal hormones
* Mammographic abnormality consistent with any type of incident breast cancer necessitating a diagnostic biopsy (BIRAD IV(b), (c) or V) will be sufficient to draw baseline LFT and complete screening questionnaire. Unless the biopsy confirms incident breast cancer, such subjects will not be included in further research interventions and they will not serve as EGCG treated or control subjects.
* Diagnosed with incident breast cancer on the diagnostic biopsy is required for inclusion in the EGCG or control treatment groups.
* Non-green tea drinker (less than monthly) - this criteria does not apply to black tea or herbal tea
* Provided written informed consent

Exclusion Criteria:

* Green tea drinker (once per month or more)
* History of breast cancer or other cancer including a prior diagnosis of any type of incident breast cancer.
* Known allergy to tea
* Abnormal liver enzymes (plus or minus 10% of the normal ranges).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-05-07 (Actual); Primary Completion 2010-12-14 (Actual); Study Completion 2016-06-06 (Actual)

PRIMARY OUTCOMES:
level of reduction in proliferation or increase in apoptosis in association with short-term EGCG | At surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wu, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States